CLINICAL TRIAL: NCT02790073
Title: Phase 2 Open Label Single Arm Repeat Dose Study to Assess the Effect of SNF472 on Wound Healing in Uraemic Calciphylaxis Patients
Brief Title: Phase 2 Study With SNF472 in Calciphylaxis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanifit Therapeutics S. A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNFCT2015_04
Record Dates: First submitted 2016-05-25; First posted 2016-06-03 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Calciphylaxis; Calcific Uremic Arteriolopathy
Keywords: Calciphylaxis; Calcific Uremic Arteriolopathy; Dialysis; End Stage Renal Disease; Rare disease (ORPHA280062); Calcification; Calcium Metabolism Disorders; Calcinosis; Metabolic Diseases
MeSH Terms: conditions — Calciphylaxis; Kidney Failure, Chronic; Rare Diseases; Calcinosis; Calcium Metabolism Disorders; Metabolic Diseases | interventions — SNF472

ARMS (1):
- SNF472 (Other): SNF472 for calciphylaxis
  Interventions: Drug: SNF472

INTERVENTIONS:
Drug: SNF472 — SNF472 for calciphylaxis

SUMMARY:
To evaluate the effect of SNF472 on top of standard of care on promoting wound healing and other parameters of therapeutic response in haemodialysis patients with calciphylaxis (calcific uraemic arteriolopathy, CUA).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with either newly diagnosed CUA OR recurrent CUA that has been dormant with no skin lesion involvement for at least 90 days from study start (new or recurrent diagnosis must be made within 5 weeks of study start)
2. Patients who signed the written informed consent to participate in this clinical trial (prior to any clinical trial-related procedures being performed), after reading the Patient Information Sheet and Informed Consent Form (ICF), and who had the opportunity to discuss the clinical trial with the Investigator or designee
3. Males or females aged ≥18
4. Patients on maintenance haemodialysis (HD)
5. Patients with at least a minimum level of pain on Visual Analog Scale (VAS) scale or on pain-killers stronger than non-steroidal anti-inflammatory drugs (NSAIDs)
6. Females of child-bearing potential should use a highly effective contraceptive measure throughout the study and have a negative serum pregnancy test at entry. Male patients having sexual relationship in which pregnancy can occur should take adequate contraceptive precautions (wear a condom)

Exclusion Criteria:

1. Body weight above 150 kg
2. BMI >35 and central(abdominal) ulcers
3. History of bisphosphonate treatment within 12 months before entering into the study
4. Severely ill patients without reasonable expectation of survival for > 6 months according to the treating physician
5. Patients with scheduled parathyroidectomy during the run-in or study period
6. Female patients who are either intending to get pregnant or are undergoing treatment to get pregnant, as well as breast-feeding females
7. Participation in another clinical trial with an experimental drug within 90 days prior the inclusion
8. Any psychological, emotional problems, any disorders or resultant therapy that is likely to invalidate informed consent, or limit the ability of the patient to comply with the Clinical Trial Protocol requirements
9. Patients who, in the opinion of the Investigator, are considered unsuitable for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Brandenburg, Principal Investigator — RWTH Aachen University
Locations (3):
- United States (2):
  - Fresenius Medical Services, Waltham, Massachusetts
  - Davita Clinical Research, Minneapolis, Minnesota
- Salford Royal Hospital, Salford, United Kingdom

REFERENCES:
- See also: USA FDA resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: Drug Information available for: SNF472 — http://www.sanifit.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNF472
Started | 14
Completed | 11
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal from HD | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | SNF472
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Wound Healing
Description: Absolute change in Bates-Jensen Wound Assessment (BWAT) total score between baseline (Week 1) and Week 12 for the primary lesion (the largest one).
  The Bates-Jensen Wound Assessment (BWAT) is a standardized tool for quantitative assessment of wound healing that includes the 13 items listed below.
  * Size
  * Depth
  * Edges
  * Undermining or pockets
  * Necrotic tissue type
  * Necrotic tissue amount
  * Exudate type
  * Exudate amount
  * Surrounding skin color
  * Peripheral tissue edema
  * Peripheral tissue induration
  * Granulation tissue
  * Epithelialization
  Each item was rated on a scale of 1 (best) to 5 (worst). The Bates-Jensen Wound Assessment (BWAT) total score is the sum of the individual items with a possible range of 13 (best) to 65 (worst).
Time Frame: 12 weeks
Population: Subjects who received at least 1 dose of SNF472 and had at least 1 postbaseline efficacy measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SNF472
Number analyzed (Participants) | 14
units on a scale | -8.1 (8.5)
Statistical Analysis 1: Comparison: SNF472; Test type: Other — Within group comparison vs baseline; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Wound Pain
Description: Absolute change from baseline (Week 1) and Week 12 in the Pain Visual Analogue Scale (VAS) Score.
  The Pain Visual Analogue Scale (VAS) Score is a horizontal line, 100 mm in length, anchored by word descriptors at each end. The subject marked the point on the line that represented his/her perception of his/her current pain status. The Pain Visual Analogue Scale (VAS) Score was determined by measuring in millimeters from the left hand end of the line (no pain) to the point that the subject marked. The Pain Visual Analogue Scale (VAS) Score range 0 (best) to 100 (Worst).
Time Frame: 12 weeks
Population: Subjects who received at least 1 dose of SNF472 and had at least 1 postbaseline efficacy measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SNF472
Number analyzed (Participants) | 14
units on a scale | -23.6 (30.0)
Statistical Analysis 1: Comparison: SNF472; Test type: Other — Within group comparison vs baseline; p = 0.015, t-test, 2 sided

3. Secondary Outcome: Wound-QoL Global Score
Description: Absolute change from baseline (Week 1) and Week 12 in the Wound-QoL global score.
  The Wound-QoL questionnaire measures the disease-specific, health related QoL of patients with chronic wounds. It consists of 17 items on impairments that are assessed in retrospect to the preceding 7 days and rated on a 0 (best) to 4 (worse) scale with possible responses from "not at all" to "very much". The total score is the average of the 17 responses.
Time Frame: 12 weeks
Population: Subjects who received at least 1 dose of SNF472 and had at least 1 postbaseline efficacy measurement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SNF472
Number analyzed (Participants) | 14
units on a scale | -0.9 (0.87)
Statistical Analysis 1: Comparison: SNF472; Test type: Other — Within group comparison vs baseline; p = 0.003, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | SNF472
All-Cause Mortality (participants affected / at risk) | 2/14
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNF472 (N=14)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNF472 (N=14)
Tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (2)
Peripheral swelling (General disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (6)
Electrocardiogram QT prolonged (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral oedema (General disorders) | 1 (1)
Cellulitis (Investigations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (5)
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT02790073/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT02790073/SAP_001.pdf